CLINICAL TRIAL: NCT04956796
Title: Effect of Airway Video Library on Intubation in Novices
Status: Withdrawn | Type: Observational
Why Stopped: PI left the institution
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00012340
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Anesthesia; Anesthesia Intubation Complication
Keywords: Intubation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: At the beginning of Phase 1, participants from Group A will be exposed to the video airway library in addition to the conventional airway training. At the beginning of Phase 2, participants will continue with conventional airway training only. Each phase will last for 1 month.
  Interventions: Behavioral: Airway Video Library Training; Behavioral: Conventional Airway Training
- Group B: At the beginning of Phase 1, participants from Group B will be exposed to the conventional airway training only. At the beginning of Phase 2, the participants in Group B will be exposed to the video airway library. Each phase will last for 1 month.
  Interventions: Behavioral: Airway Video Library Training; Behavioral: Conventional Airway Training

INTERVENTIONS:
Behavioral: Airway Video Library Training — A video airway library consisting of real-life clinical videos of laryngoscopy and endotracheal intubation was developed by the study investigators. This library consists of video clips of normal and easy airways, pediatric airways as well as pathological or difficult airways that is devoid of patient identifying data. The participants of the study group will be exposed to the video library by two learning sessions. Each learning session consists of 1 hour of interactive & immersive learning of 30 airway videos. At the end of the session, the participants will be oriented to the airway and identify key airway structures, learn to troubleshoot and navigate difficult anatomy, optimize visualization, and use accessory airway equipment.
Behavioral: Conventional Airway Training — The endotracheal intubation training Anesthesiology students currently receive routinely as part of their education.

SUMMARY:
Endotracheal intubation requires significant training and expertise. This experience can be quite stressful for novice users. To accelerate the learning curve of newly enrolled trainees to assess and secure airway, the investigators propose supplementing current training techniques with access to an airway video library consisting of real- life clinical videos of airway and endotracheal intubations.

DETAILED DESCRIPTION:
Timely and correctly performed endotracheal intubation is important. It can be stressful especially among beginners and requires significant expertise. Studies suggest that endotracheal intubation success rates are below 50% for the first 10 intubations among novices and the learning curve of laryngoscopy does not plateau above a 90% success rate until a mean of 57 attempts. Although simulation, which is currently the mainstay of training for airway management help orient a novice user, it is siloed from the actual experience. Endotracheal intubation requires significant training and expertise. This experience can be quite stressful for novice users. To accelerate the learning curve of newly enrolled trainees to assess and secure airway, the investigators propose supplementing current training techniques with access to an airway video library consisting of real- life clinical videos of airway and endotracheal intubations.

ELIGIBILITY:
Inclusion Criteria:

* Incoming anesthesia resident (CA-1 year)

Exclusion Criteria:

* Participants with prior experience of more than 60 intubations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All the anesthesia residents employed by the University of Minnesota (UMMC) and part of the Fairview system comprise the study population. The clinic/hospitals these residents (CA-1 year) are affiliated with include University of Minnesota Medical Center East and West Bank and VA Minneapolis.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Number of Attempts to Successful Intubation | 2 months
  Intubation success rate will be reported in number of attempts, where lower values equate to greater success. Supervising staff report success rates.
Time for Successful Intubation | 2 months
  Time to successful intubation will be measured in seconds as reported by supervising staff.
Difficulty Level of Intubation as Assessed by Intubation Difficulty Scale | 2 months
  The supervising staff fills out a questionnaire that assesses the technical skill of laryngoscopy and the complexity of intubation as per the Intubation Difficulty Scale (IDS). Those with and without exposure to the video library will be compared. The IDS is a sum of 7 parameters. The sum value of 0 indicates easy intubation, 1-5 indicates slight difficulty, and values greater than 5 indicate moderate to high difficulty.

SECONDARY OUTCOMES:
Stress Level as Assessed by Ottawa Mood Scales | 2 months
  The participant fills in the Stress Scale item of the Ottawa Mood Scales with Likert scale response to reflect the stress they experienced surrounding endotracheal intubation. The scale ranges from 0 to 10, where higher scores indicate greater stress. Those with and without exposure to the video library will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Tjorvi Perry, MD, MMSc, Principal Investigator — Univeristy of Minnesota Medical School Department of Anesthesiology
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No